CLINICAL TRIAL: NCT02797379
Title: The Development of a Psychoeducation Tool to Manage Anxiety in People With Autism Spectrum Disorders: the Managing Anxiety iN Autism GuidE (MANAGE)
Brief Title: The Development of a Psychoeducational Tool to Manage Anxiety in People With Autism Spectrum Disorders
Acronym: MANAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other); Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200774
Record Dates: First submitted 2016-05-24; First posted 2016-06-13 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2016-09

CONDITIONS: Autism Spectrum Disorders; Anxiety
Keywords: Psychoeducation; Self-help
MeSH Terms: conditions — Autism Spectrum Disorder; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate start (Other): This group receive the intervention (psychoeducation guide) immediately following baseline assessment and are assessed 4 and 8 weeks later.
  Interventions: Other: Psychoeducation
- Delayed start (Other): This group do not receive the intervention for 4 weeks. They are assessed after the wait period (4 weeks) and again after 4 weeks of having the intervention (psychoeducation guide) at week 8.
  Interventions: Other: Psychoeducation

INTERVENTIONS:
Other: Psychoeducation — The intervention is focused on psychoeducation. Four psychoeducation guides will be available: parent/caregiver, adult with ASD, adolescent with ASD, and child with ASD. The guides introduce the concept of anxiety and how it presents in individuals with ASD, different anxiety triggers, strategies that can be used to manage anxiety, and an introduction to specific anxiety disorders. Level of detail, language and presentation of content will vary across the guides to be appropriate for the functioning level of the readers.
  Other Names: Self-help guide

SUMMARY:
The purpose of this pilot intervention trial is to assess the efficacy of newly developed psychoeducation guides designed to manage anxiety in Autism Spectrum Disorder (ASD) by recruiting 30 participants with ASD and high levels of anxiety along with their parent/caregivers who both receive a version of the psychoeducation guide.

DETAILED DESCRIPTION:
ASDs have a devastating impact on adaptive function; current UK lifetime costs of supporting a person with an ASD, along with the opportunity costs of lost productivity, are estimated at £0.8-1.2 million per year (Knapp, Romeo, & Beecham, 2009). The impact of having an anxiety disorder has also been shown to affect an individual's quality of life and functioning over and above physical illness, major depression and socioeconomic factors (Stein et al., 2010). Around 40% of individuals with ASD will also have anxiety symptoms, and treatment for additional mental health problems is also costly. Early work using clinical therapies with individuals with ASD such as modified CBT indicate that the anxious symptoms which co-occur with ASD can be modified and improvements to the anxiety recorded although further work is needed. Therefore, focussing on interventions for individuals with ASD and anxiety may be very beneficial. However, not all individuals with ASD that also present with anxiety will require face to face therapy, therefore, psychoeducation could provide an effective and cost-effective way of improving mental health in ASD through self-help strategies. This could lead to improved outcomes for individuals and less burden on the clinical services supporting these families.

The intervention is focused on psychoeducation. Four psychoeducation guides will be available: parent/caregiver, adult with ASD, adolescent with ASD, and child with ASD. Participants and their parents/caregivers will be give guides to read in their own time over a 4 week period. The guides will be designed to improve participant's and their parent/caregiver's knowledge of anxiety in ASD. The guides introduce the concept of anxiety and how it presents in individuals with ASD, different anxiety triggers, strategies that can be used to manage anxiety, and an introduction to specific anxiety disorders. Level of detail, language and presentation of content will vary across the guides to be appropriate for the functioning level of the readers.

The aim of this study is to recruit 30 participants with autism spectrum disorder (ASD) and high levels of anxiety (aged 8-25 years) and their parent/caregiver into a pilot trial of a psychoeducation intervention. Participants will be recruited through clinical services in South London and the Maudsley (SLaM) and Guy's and St Thomas' (GSTT) NHS trusts through the patient consent to contact register (C4C) in SLaM and via referral from clinical care co-ordinators in the clinics in each trust. Additional participants may be recruited from non-clinical sources such as research recruitment lists held by autism charities or advertisements, including local newsletters, social media sites, emails or letters.

This is a pilot efficacy trial of newly developed psychoeducation guides employing a randomized, parallel-arm, intention to treat design with a 4 week intervention. Participant families will be randomly allocated (1:1) to either an immediate or a delayed start group to allow measurement of anxiety symptoms over a one month period with and without the psychoeducation guide. This design helps to control for the effects of attention (anxiety may show a large placebo response) while allowing all participants access to the intervention.

The aim is to improve participants' and their parent/caregivers' knowledge of the presentation of anxiety in ASD and their confidence in using simple strategies in its management. The primary outcome is improvement of participant and parent/caregiver understanding of the presentation and simple management strategies for anxiety in ASD. Secondary outcomes include improvement in anxiety symptoms and confidence in managing anxiety, feedback on acceptability, usefulness and appropriateness of the guide.

The trial analyses will be intention-to treat. Missing data will be imputed. The primary analysis will compare the groups randomized to immediate vs delayed treatment 4 weeks post randomisation when the immediate start group will have had the guide for 4 weeks and the delayed start group will have been on a "waiting list" for 4 weeks, this controls for attention and spontaneous improvement. The investigators will then check the two groups for comparability at pre-intervention time point (Time 1). If the two groups show similar baselines levels and magnitude of change in knowledge and symptom severity post intervention, they will be combined to gain a further estimate of the treatment effect. Both the knowledge/confidence measure and measure of anxiety symptoms, will be treated as continuous variables. Linear regression models will include baseline severity and randomisation group as predictors. The primary focus will be on parent-carer response but if sample sizes are sufficient, separate, parallel analyses will use data from individuals with ASD.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of ASD.
* Elevated levels of anxiety according to baseline questionnaire measure (Screen for Anxiety Related Disorders; SCARED)
* Have a parent/caregiver who is knowledgeable about participant's mental state and everyday activities and who can facilitate their use of the psychoeducation guide
* Mental age of 8 years or older, the lowest age recommended to complete the standardised measure of anxiety.

Exclusion Criteria:

* Participants or consultees, where relevant, who are unwilling to participate
* Participants who do not have a reasonable level of English. This is because a reasonable level of English will be required to engage with the guide, which is presently written in English and the questionnaires and/or interview questions about the guide. With younger participants with ASD using the materials, English should be the language used at home and school.
* Participants with any significant safeguarding concerns or involvement with court proceedings.
* Participants who are due to commence or have a major change in psychological or pharmacological treatment for their anxiety at a similar time to being given the psychoeducation guide.

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Knowledge about anxiety in ASD | 4 weeks of using the guide
  The primary objective is to improve the participants' and their parent/caregivers' knowledge of the presentation of anxiety in ASD management from pre- to post-intervention. This will be measured after 4 weeks of using the psychoeducation guide (this will be 4 weeks post-randomisation for the immediate start group and 8 weeks post-randomisation for the delayed start group).

SECONDARY OUTCOMES:
Anxiety symptoms | 4 weeks of using the guide
  One secondary aim will be to determine whether use of the guide leads to a decrease in reported anxiety symptoms in the participant and their impact on everyday life. This will be measured pre and post intervention with the Screen for Anxiety Related Disorders.
Acceptability, usefulness and appropriateness of the guide | 4 weeks of using the guide
  In providing the participant and/or their parent/caregiver with the psychoeducation guide the research team will also seek feedback on acceptability, usefulness and appropriateness of the guide for each participant. This will be measured using newly developed feedback questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Simonoff, MD, Principal Investigator — King's College London
Locations (2):
- United Kingdom (2):
  - South London and the Maudsley, London
  - Guy's and St Thomas' NHS trust, London

IPD SHARING:
Plan to Share IPD: No